CLINICAL TRIAL: NCT01740180
Title: Cortico-saving Treatments Proposed for CLIPPERS (Chronic Lymphocytic Inflammation With Pontine Perivascular Responsive to Steroids): a First Cohort
Brief Title: Cortico-saving Treatments Proposed for CLIPPERS: a First Cohort
Status: Terminated | Type: Observational
Why Stopped: No recruitment
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2012/GT; Taieb Cohorte CLIPPERS (Other: BESPIM, Nîmes University Hospital)
Record Dates: First submitted 2012-11-30; First posted 2012-12-04 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2018-01

CONDITIONS: CLIPPERS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CLIPPERS patients: The population concerned by this study consists of patients diagnosed according to CLIPPERS criteria (see inclusion and exclusion criteria).
  Intervention: Data entry
  Interventions: Other: Data entry

INTERVENTIONS:
Other: Data entry — This cohort describes the basic information about the patients (age, sex, weight, height, background) as well as acts required, treatment and results of imaging studies.
  These data are extracted from patient records by each participating center and collected in an e-CRF.

SUMMARY:
The primary objective of this study is to collect information about how CLIPPERS patients are currently being treated in France.

DETAILED DESCRIPTION:
This is an observational study. Data will be prospectively collected, starting with a detailed baseline description of disease and treatment status, followed by updates everything six months for the next three years.

ELIGIBILITY:
Inclusion Criteria:

* Patient correctly informed about the study
* Symptoms and/or clinical signs indicating that the brain stem is affected
* MRI shows punctate gadolinium highlights and/or curvilinear bridge and/or middle cerebellar peduncles
* Clinical and radiological cortico sensitivity
* If a cerebral biopsy has been performed, presence of a lymphocytic, histiocytic or lympho-hysticytic infiltrate

Exclusion Criteria:

* symptoms and/or clinical signs indicating impairment other than the central nervous system
* Cortical impairment present on MRI, microbleeds, stenosis on magnetic resonance angiography, or pacchymeningitis
* Presence of other diseases that could explain such clinical and radiological signs (see inclusion criteria)
* If a cerebral biopsy has been performed, presence of signs of malignancy (eg, clonal proliferation, cellular atypia), vasculitis, granuloma, or demyelination

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population concerned by this study consists of patients diagnosed according to CLIPPERS criteria (see inclusion and exclusion criteria).
  Patients will be recruited from referral centers throughout France. We also intend to communicate with all multiple sclerosis networks (French League against Multiple Sclerosis) to facilitate the detection of new cases.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2015-03-25 (Actual); Primary Completion 2016-03-25 (Actual); Study Completion 2016-03-25 (Actual)

PRIMARY OUTCOMES:
Presence/absence of cortico-sparing treatments | baseline to 3 years

SECONDARY OUTCOMES:
Presence/absence of allergies | Baseline (day 0)
  + description
Complete description of all treatments being taken | Baseline (day 0)
CLIPPERS relapse severity | Baseline (day 0)
  The rhythm and severity of relapses.
Relapse-free interval rhythm | Baseline (day 0)
Weight (kg) | Baseline (day 0)
Presence/absence of vascular risk factors | Baseline (Day 0)
Number of relapses in the past 6 months while taking >= 20 mg/ day corticoids | Baseline (day 0)
Presence/absence of allergies | 6 months
  + description
Presence/absence of allergies | 12 months
  + description
Presence/absence of allergies | 18 months
  + description
Presence/absence of allergies | 21 months
  + description
Presence/absence of allergies | 24 months
  + description
Presence/absence of allergies | 30 months
  + description
Presence/absence of allergies | 36 months
  + description
Complete description of all treatments being taken | 6 months
Complete description of all treatments being taken | 12 months
Complete description of all treatments being taken | 18 months
Complete description of all treatments being taken | 21 months
Complete description of all treatments being taken | 24 months
Complete description of all treatments being taken | 30 months
Complete description of all treatments being taken | 36 months
CLIPPERS relapse severity | 6 months
  The rhythm and severity of relapses.
CLIPPERS relapse severity | 12 months
  The rhythm and severity of relapses.
CLIPPERS relapse severity | 18 months
  The rhythm and severity of relapses.
CLIPPERS relapse severity | 21 months
  The rhythm and severity of relapses.
CLIPPERS relapse severity | 24 months
  The rhythm and severity of relapses.
CLIPPERS relapse severity | 30 months
  The rhythm and severity of relapses.
CLIPPERS relapse severity | 36 months
  The rhythm and severity of relapses.
Relapse-free interval rhythm | 6 months
Relapse-free interval rhythm | 12 months
Relapse-free interval rhythm | 18 months
Relapse-free interval rhythm | 21 months
Relapse-free interval rhythm | 24 months
Relapse-free interval rhythm | 30 months
Relapse-free interval rhythm | 36 months
Weight (kg) | 6 months
Weight (kg) | 12 months
Weight (kg) | 18 months
Weight (kg) | 21 months
Weight (kg) | 24 months
Weight (kg) | 30 months
Weight (kg) | 36 months
Presence/absence of vascular risk factors | 6 months
Presence/absence of vascular risk factors | 12 months
Presence/absence of vascular risk factors | 18 months
Presence/absence of vascular risk factors | 21 months
Presence/absence of vascular risk factors | 24 months
Presence/absence of vascular risk factors | 30 months
Presence/absence of vascular risk factors | 36 months
Number of relapses in the past 6 months while taking >= 20 mg/ day corticoids | 6 months
Number of relapses in the past 6 months while taking >= 20 mg/ day corticoids | 12 months
Number of relapses in the past 6 months while taking >= 20 mg/ day corticoids | 18 months
Number of relapses in the past 6 months while taking >= 20 mg/ day corticoids | 21 months
Number of relapses in the past 6 months while taking >= 20 mg/ day corticoids | 24 months
Number of relapses in the past 6 months while taking >= 20 mg/ day corticoids | 30 months
Number of relapses in the past 6 months while taking >= 20 mg/ day corticoids | 36 months

OTHER OUTCOMES:
Family history of auto-immune disease | Baseline
Height (cm) | Baseline (day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Taieb, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (11):
- France (11):
  - CHU de Bordeaux - Groupe Hospitalier Pellegrin, Bordeaux
  - CH de Dax - Côte d'Argent, Dax
  - CHU de Limoges - Hôpital Dupuytren, Limoges
  - APHM - Hôpital La Timone Adultes, Marseille
  - CHU de Montpellier - Hôpital Saint-Eloi, Montpellier
  - CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes
  - CHU de Rouen - Hôpital Charles Nicolle, Rouen
  - CHRU de Strasbourg - Hôpital Civil, Strasbourg
  - CHRU de Toulouse - Hôpital de Rangueil, Toulouse
  - CHRU de Toulouse - Hôpital Purpan, Toulouse
  - CHRU de Tours - Hôpital Bretonneau, Tours